CLINICAL TRIAL: NCT03581526
Title: Psychological and Behavioral Change Before and After General Anesthesia in Preschool Children: Preliminary Study
Brief Title: Mood Change After General Anesthesia in Children
Status: Completed | Type: Observational
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Other Study IDs: DCMC#4
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia, General; Psychology, Child; Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most drugs used in general anesthesia work on various receptors in the human brain, causing unconsciousness, loss of memory, and loss of reflection of the autonomic nervous system. After the anesthesia, baseline physiological function will be attained by administration of some reversal drugs or as the time goes by. In this process, various side effects may occur.

Emergence delirium (ED) is a representative behavioral disturbance after general anesthesia in children and that can cause several problems during the recovery period. Previous studies found that ED and postoperative behavioral problems might be connected. Preschoolers are the most vulnerable group in developing ED after general anesthesia, however, it is difficult to evaluate the psychiatric problems at this age.

The Child Behavior Checklist (CBCL) 1.5-5 is an internationally well-known standardized tool for assessment of developmental psychopathology, consisted of 99 problem items. Items are categorized as following syndrome scales: Emotionally reactive, Anxious/Depressed, Somatic complaints, Withdrawn, Attention problems, Aggressive behavior, and sleep problems.

In this study, the investigators would observe the behavioral and emotional changes of the child using the CBCL 1.5-5 between before and after the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 7 years of American Society of Anesthesiologists physical status (ASA PS) I or II who are planned to receive surgery under general anesthesia

Exclusion Criteria:

* If the guardian and the subject are difficult to evaluate normally due to language barriers/language disorders/delay or autistic disorder
* with developmental delay, neurological disorders or psychiatric diseases associated with symptoms of agitation, anxiety, attention deficit, sleep disturbances, etc
* refusal of consent
* Any visual or auditory problems of the primary responder of CBCL
* recently received psychiatric medication or sleep supplements
* Recent history (within a month) of received general anesthesia or surgery

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged between 2 and 7 years
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Change of T-score of total score of child behavior checklist 1.5-5 (CBCL 1.5-5) | before anesthesia induction and 1 week after the surgery
  T-score is the scale in order to indicate the relative position within the whole group that has been standardized, the average and standard deviation of the percentile distribution obtained through the origin sum of score. The CBCL 1.5-5 included 99 questions that describe specific kinds of behavioral and emotional problems for preschool children. Questions are scored on syndrome scales designated as emotionally reactive, anxious/depressed, somatic complaints, withdrawn, attention problems, aggressive behavior, and sleep problems. Higher scores mean great behavioral disturbances.
Change of T-score of each internalizing problems | before anesthesia induction and 1 week after the surgery
  T-score is the scale in order to indicate the relative position within the whole group that has been standardized, the average and standard deviation of the percentile distribution obtained through the origin sum of score. Internalizing problems are consisted of following 4 categories : emotionally reactive, withdrawn, somatic complaints, and anxious/depressed.
  The subjects are asked to answer the questions with a 3 point scale:
  0 for not true of the child; 1 for somewhat or sometimes true, and 2 for very true of often true. The scores for problems were calculated according to the CBCL manuals. Higher scores mean great behavioral disturbances.
Change of T-score of each externalizing problems | before anesthesia induction and 1 week after the surgery
  T-score is the scale in order to indicate the relative position within the whole group that has been standardized, the average and standard deviation of the percentile distribution obtained through the origin sum of score.
  Externalizing problems are consisted of following 2 categories : Attention problems and aggressive behavior.
  The subjects are asked to answer the questions with a 3 point scale:
  0 for not true of the child; 1 for somewhat or sometimes true, and 2 for very true of often true. The scores for problems were calculated according to the CBCL manuals. Higher scores mean great behavioral disturbances.
Change of T-score of sleep problems | before anesthesia induction and 1 week after the surgery
  T-score is the scale in order to indicate the relative position within the whole group that has been standardized, the average and standard deviation of the percentile distribution obtained through the origin sum of score. The subjects are asked to answer the questions with a 3 point scale:
  0 for not true of the child; 1 for somewhat or sometimes true, and 2 for very true of often true. The scores for problems were calculated according to the CBCL manuals. Higher scores mean great behavioral disturbances.
Emergence Delirium (ED) | Approximately during 60 min after PACU admission
  Whether ED is occurs during PACU stay in children. The determination of ED was made using parameters PAED >12 and Watcha >2.

SECONDARY OUTCOMES:
modified Yale preoperative anxiety score (mYPAS) | before anesthesia induction (about 30 min before the surgery)
  mYPAS is the assessment tool for measure the anxiety before induction. Higher score indicates higher anxiety.
PAED score during PACU stay | During 60 min after PACU admission
  On arrival at post-anesthesia care unit (PACU) and every 10 min from then, patients were checked PAED. The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.
Watcha scale on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  On arrival and 10, 20, and 30 min after PACU admission, patients were checked Watcha scale as following 4-point scale
  calm crying, but can be consoled Crying, cannot be consoled Agitated and thrashing around
FLACC score on initial, 10, 20, and 30 min | During 60 minutes after PACU admission
  Face, legs, activity, cry, and consolability (FLACC) score is checked every 10min after PACU admission
Postoperative adverse event | During 60 minutes after the surgery
  After the end of surgery, postoperative adverse events (such as postoperative dizziness, sore throat, abdominal pain, breath holding, coughing, desaturation, laryngospasm, and bronchospasm) are checked during emergence period and PACU stay.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, PhD, Study Chair — Assistant professor; JongHae Kim, MD, Study Director — Associate professor; Sooyeon Kim, MD, Principal Investigator — Fellow
Locations (2):
- South Korea (2):
  - Daegu Catholic University Medical Center, Daegu
  - Hanyang University medical center, Seoul